CLINICAL TRIAL: NCT03609645
Title: Optimization of Analgesia for Hip Fracture: Femoral and Obturator Articular Branch Block vs. Fascia Iliaca Block. A Double-blind, Randomized- Controlled Trial.
Brief Title: Optimization of Analgesia for Hip Fracture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-6067
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-07

CONDITIONS: Hip Fractures
Keywords: Fascia Iliaca Block; Femoral and Obturator Articular Branch Block
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomized prospective study involving patients with hip fracture who are undergoing surgical fixation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An unblinded study personnel not directly involved in patient care will prepare all study drugs. The anesthesiologist, patient, surgeon and the investigator collecting outcome data will be unaware of study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca block (FIB) (Active Comparator): Group will receive Fascia iliaca block (FIB) with local anesthetic and femoral articular branch block (FAB) with normal saline (Placebo).
  Interventions: Procedure: Fascia iliaca block
- Femoral articular branches block(FAB) (Experimental): Group will receive Fascia iliaca block (FIB) with normal saline (Placebo) and Femoral AON articular branch block (FAB) with local anesthetic.
  Interventions: Procedure: Femoral articular branches block(FAB)

INTERVENTIONS:
Procedure: Fascia iliaca block — FIB Placebo Block: 20mL of Normal Saline Active drug: 20mL of 0.25% Bupivacaine with epinephrine (1:400, 000)
  FAB block Placebo Block: 20mL of Normal Saline Active Drug: 20mL of 0.25% Bupivacaine with epinephrine (1:400,000)
  Arms: Fascia iliaca block (FIB)
Procedure: Femoral articular branches block(FAB) — FIB Placebo Block: 20mL of Normal Saline Active drug: 20mL of 0.25% Bupivacaine with epinephrine (1:400, 000)
  FAB block Placebo Block: 20mL of Normal Saline Active Drug: 20mL of 0.25% Bupivacaine with epinephrine (1:400,000)
  Arms: Femoral articular branches block(FAB)

SUMMARY:
Hip Fracture is a common orthopedic emergency in elderly people, which causes moderate to severe pain. Until now, different methods of pain treatment have been used, including pain-killer medication, which given in to the vein, and a nerve block.. A nerve block is the defined as injection of a freezing/numbing medication (local anesthetic) around the nerve area in order to stop pain.

Painkiller medications by themselves are not enough to stop pain, especially the pain that start with movement.

At the Toronto Western hospital, patients with hip fracture will generally receive a fascia iliac block (FIB) within 24 hours of hospital admission as a standard of care.

Fascia iliaca block is a nerve block done by injecting local anestheticat the level of the groin. This done to provide pain relief and is done either in the emergency room or in the inpatient area.

Studies have shown that nerves supplying other areas in the hip may be blocked to relive hip pain fracture.

Additional to this method, there is a newer type of nerve block, called the femoral articular branch block (FAB) that aim to block the nerves supplying the hip joint.

This new block has been described based on better understanding of the anatomy of the nerves that control hip pain. This block consists on an injection in the groin at a similar location as the Fascia iliaca block except that the needle has to go slightly deeper (by a few centimeters) to reach a better target.

Based on the current understanding on anatomy it is possible that this new technique may provide better pain control than a Fascia Iliaca Block.

The purpose of the study is to investigate the degree of pain relief achieved by the two different nerve block techniques: 1) Fascia iliaca block (FIB) and 2) Femoral and AON articular branches block (FAB).

DETAILED DESCRIPTION:
The anterior hip joint is innervated by articular branches from the femoral nerve (FN), the obturator nerve (ON) and the accessory obturator nerve (AON). The posterior and inferior parts of the hip joint capsule are innervated by the sacral plexus via a) the sciatic nerve, b) the sciatic branch to the quadratus femoris muscle and c) the superior gluteal nerves. Gerhardt et al showed that nociceptive fibers are predominantly present in the anterior and superolateral parts of the joint capsule, suggesting that the femoral and obturator nerves should be the most important nerves to target for hip analgesia.

The 3-in-1 block and FIB are currently used to provide hip analgesia. However, recent MRI imaging studies have shown that proximal local anesthetic spread was not consistent following a 3-in-1 block and did not consistently cover the obturator nerve. Similar findings were reported for the FIB.

A recent study on the innervation of the anterior hip revealed the relevant landmarks for the articular branches of the FN, AON and ON. This study found that high branches of femoral nerve, which were given off superior to the inguinal ligament, play a greater role in the anterior hip innervation than previously reported. These high articular branches of the FN and AON are consistently found between anterior inferior iliac spine (AIIS) and iliopubic eminence (IPE). With the help of ultrasound imaging, these landmarks can be identifiable and it is possible to target them directly in order to provide hip analgesia.

These recent data suggests that blocking these branches as they course deep to the iliopsoas muscle should result in superior hip joint analgesia compared to a FIB since the local anesthetic spread from a FIB is neither proximal nor deep enough to cover these articular branches consistently. Real-time ultrasound can help identify these proximal FN and AON branches using the anterior inferior iliac spine and the iliopubic eminence as landmarks.

The overall aim of this study is to determine in a prospective, randomized, double blind manner, the analgesic profile associated with two different regional anesthetic techniques: (1) FIB and (2) Femoral articular branches (FAB) block.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I-III
* 60 years old or older
* BMI 18-40
* Scheduled for hip fracture surgical fixation

Exclusion Criteria:

* Bilateral hip fracture
* Lack of mental ability to provide informed consent
* Pre-existing neuropathic pain or sensory disorders of the surgical limb
* Contraindication to regional anesthesia (Intolerance to the study drugs, bleeding diathesis, coagulopathy, malignancy or infection at the site of the block)
* Chronic opioid use defined as >30 mg of daily oral morphine equivalents

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic pain score | 60 minutes after the block procedure
  Pain scores will be assessed with an 11-point verbal numeric rating scale (NSR) where 0 is "no pain" and 10 is "the worst pain imaginable" and dynamic pain will be assessed with 15 degrees straight leg raise.
  The 15 degrees straight leg raise is a safe and standardized test to evaluate dynamic pain in hip fracture patients and has been used in a previous study.

SECONDARY OUTCOMES:
Rest pain score | 30, 60, 120 and 180 minutes post-block
  Pain scores will be assessed with an 11-point verbal numeric rating scale (NSR) where 0 is "no pain" and 10 is "the worst pain imaginable" and dynamic pain will be assessed.
Dynamic pain score | 30, 120 and 180 minutes post-block
  Pain scores will be assessed with an 11-point verbal numeric rating scale (NSR) where 0 is "no pain" and 10 is "the worst pain imaginable" and dynamic pain will be assessed with 15 degrees straight leg raise.
Cumulative systemic opioid consumption | 1 hour, 3 hours and 24 hours after the block procedure
  oral morphine mg equivalents
Requirement "rescue" intravenous patient controlled analgesia (IV PCA) | within first 24 hours after the block procedure
  If oral pain medication and block is not enough patient can get IV PCA.We will be recording requirement of IV PCA anytime in the first 24 hours after the block procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Peng, MD, Principal Investigator — University Health Network-Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada